CLINICAL TRIAL: NCT05931029
Title: Study of the Therapeutic Effects of Naohuan Dan and Idebenone in Treating Mild Cognitive Impairment With Kidney Deficiency and Phlegm Stasis
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-332-01
Record Dates: First submitted 2023-06-08; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — idebenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The control group: The control group received Idebenone orally, at a dose of 30mg per time, three times a day, after meals for 12 consecutive weeks.
  Interventions: Drug: Idebenone
- The treatmen group: The treatment group received Naohuan Dan combined with Idebenone. At a dose of one per day, delivered with warm water in the morning and evening, and taken orally for 12 consecutive weeks.
  Interventions: Drug: Naohuan Dan and Idebenone

INTERVENTIONS:
Drug: Idebenone — The control group took Idebenone orally for 12 weeks.
  Groups: The control group
Drug: Naohuan Dan and Idebenone — The treatment group took Naohuan Dan combined with Idebenone for treatment. Naohuan Dan is a granular preparation taken once a day, while Idebenone is a tablet taken three times a day for a total of 12 weeks.
  Groups: The treatmen group

SUMMARY:
This study conducted a retrospective analysis of 64 patients with mild cognitive impairment of the kidney deficiency phlegm and stasis type who underwent treatment with Naohuan Dan combined with Idebenone. The patients' cognitive function was evaluated using the Mini-Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA) before and after treatment. Daily living abilities were assessed using the Activities of Daily Living (ADL) scale, depression status was evaluated using the Geriatric Depression Scale (GDS), and the severity of Traditional Chinese Medicine (TCM) syndrome was assessed using the TCM diagnostic scale. Peripheral blood from the patients was also collected for analysis of neuron-specific enolase (NSE) and inflammatory factors. The aim was to evaluate the safety and feasibility of using Naohuan Dan combined with Idebenone for the treatment of mild cognitive impairment of the kidney deficiency phlegm and stasis type.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis in accordance with both Chinese medicine and Western medicine.
* Age between 55 and 85 years, with no gender restrictions.
* A score between 21 and 26 on the Mini-Mental State Examination (MMSE), with 1 point for primary school education.
* Willingness to participate in the study and signing of the informed consent form.

Exclusion Criteria:

* Patients with severely impaired heart, liver, kidney, or other organs functions.
* Patients with neurological diseases that affect brain function and cognitive impairment.
* Patients with severe depression or other mental illnesses.
* Patients with poor compliance or cooperation who were unable to complete the study according to the protocol.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants were selected at the Traditional Chinese Medicine's and Rehabilitation Medicine's out-patient clinic or inpatient department of Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change from the Mini-Mental State Examination scale (MMSE) at 12 weeks | The time of measurement for the scale occurred twice, with the first measurement taking place before subjects were enrolled, and the second occurring at the end of their 12-week continuous medication period. Each assessment will last for one day.
  The MMSE scale measures various cognitive domains, including orientation (10 points), memory (3 points), attention and calculation (5 points), recall ability (3 points) and language skills (9 points).
Change from the clinical efficacy at 12weeks | The time of measurement for the scale occurred twice, with the first measurement taking place before subjects were enrolled, and the second occurring at the end of their 12-week continuous medication period. Each assessment will last for one day.
  The clinical efficacy was evaluated based on the MMSE scale, and the efficacy was calculated by comparing the scores before and after the therapy. The following criteria were used to determine the efficacy: (i) Markedly effective: ≥20% improvement in MMSE score. (ii) Effective rate: ≥12% improvement in MMSE score. (iii) Ineffective: <12% improvement in MMSE score.

SECONDARY OUTCOMES:
Change from the Montreal Cognitive Assessment scale (MoCA) at 12 weeks | The time of measurement for the scale occurred twice, with the first measurement taking place before subjects were enrolled, and the second occurring at the end of their 12-week continuous medication period. Each assessment will last for one day.
  The MoCA scale is a widely used screening tool for detecting mild cognitive impairment. The total score on the MoCA scale is 30, and a score of 26 or higher is considered to indicate normal cognitive function.
Change from the Activities of Daily Living scale (ADL) at 12 weeks | The time of measurement for the scale occurred twice, with the first measurement taking place before subjects were enrolled, and the second occurring at the end of their 12-week continuous medication period. Each assessment will last for one day.
  The ADL scale is used to assess the participants' ability to perform daily living activities. The total score on the ADL scale is 100 points.
Change from the Geriatric Depression scale (GDS) at 12 weeks | The time of measurement for the scale occurred twice, with the first measurement taking place before subjects were enrolled, and the second occurring at the end of their 12-week continuous medication period. Each assessment will last for one day.
  The GDS scale is a self-report assessment tool used to detect and measure the severity of depression in older adults. The total score on the GDS scale is 30 points.
Change from the traditional Chinese medicine (TCM) syndrome score scale at 12 weeks | The time of measurement for the scale occurred twice, with the first measurement taking place before subjects were enrolled, and the second occurring at the end of their 12-week continuous medication period. Each assessment will last for one day.
  The TCM clinical symptoms of the participants were evaluated using the TCM syndrome score scale. This tool assesses the severity of specific TCM symptoms and divides them into four grades: none, mild, moderate, and severe, with 0, 2, 4, and 6 points (for main symptoms) or 0, 1, 2, and 3 points (for secondary symptoms), respectively.
Change from the Serological indicators at 12 weeks | The time of measurement for the scale occurred twice, with the first measurement taking place before subjects were enrolled, and the second occurring at the end of their 12-week continuous medication period. Each assessment will last for one day.
  Blood samples were collected from the participants before and after the therapy via cubital venipuncture. Enzyme-linked immunosorbent assay (ELISA) was used to determine the serum levels of neuron-specific enolase (NSE), interleukin-8 (IL-8) and tumor necrosis factor-alpha (TNF-α).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital，Sun Yat-sen University，Guangzhou 510300，China, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Time Frame: Starting 6 months after publication
Access Criteria: If necessary, please request all data to the email address of the person in charge：hqhui84181833@sina.com

DOCUMENTS (2):
  • Study Protocol (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05931029/Prot_000.pdf
  • Informed Consent Form: Consent Form (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT05931029/ICF_001.pdf